CLINICAL TRIAL: NCT07034950
Title: Study on the Effective Dose and Safety of Esketamine During Ultrasound-guided Hepatic Tumor Thermal Ablation Under Hilar Nerve Blockade
Brief Title: Effective Dose and Safety of Esketamine During Ultrasound-guided Hepatic Tumor Thermal Ablation
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Lijuan Yan, Scientific Research Secretary of the Anesthesiology Department, The First Affiliated Hospital of Xiamen University
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: XMFHIIT-2025SL091
Record Dates: First submitted 2025-05-29; First posted 2025-06-24 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-06

CONDITIONS: Hepatic Neoplasm; Hepatic Cancer
Keywords: hepatic hilar nerve block; Ultrasound-guided; Thermal Ablation; Esketamine; Pain
MeSH Terms: conditions — Liver Neoplasms; Pain | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: This research will be divided into two stages.
  (i) In Phase one, a prospective dose discovery study using the Dixon sequential method will be conducted, aiming to determine the median effective dose (ED50) and 95% effective dose (ED95) of esketamine during ultrasound-guided hepatic tumor thermal ablation under hilar nerve block (HHNB). The sample size is approximately 27.
  (ii) The investigators will conduct a single-center, randomized, double-blind controlled trial in Phase Two to evaluate the safety of the esketamine ED95 dose under the monitoring anesthesia care program based on the incidence of respiratory depression. The intervention group will be injected with the dose of esketamine ED95; the control group will be injected with fentanyl 1 μg∙kg-1. Both groups of patients will receive the same sedation regimen. The sample size is approximately 52.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Determine the ED50 and ED95 of esketamine by Dixon's up-and-down method (Experimental): Using Dixon's up-and-down sequential method, esketamine will be titrated intravenously from an initial 0.3 mg∙kg-1 dose with 0.02 mg∙kg-1 adjustments based on intraprocedural responses to pain (positive: purposeful somatic movement or the complaint of pain; negative: no movement or no complaint of pain). All patients will receive standardized premedication with HHNB. The titration sequence will continue until six crossover inflection points are observed.
  Interventions: Drug: Intravenous esketamine using Dixon's up-and-down sequential method
- Evaluate the safety of the dose of esketamine ED95 by the incidence of respiratory depression (Active Comparator): The intervention group will be injected with the dose of esketamine ED95; the control group will be injected with fentanyl 1 μg∙kg-1. The study at this stage will evaluate the safety of the dose of esketamine ED95 through the incidence of respiratory depression.
  Interventions: Drug: Intravenous the dose of esketamine ED95; Drug: Intravenous fentanyl 1 μg∙kg-1

INTERVENTIONS:
Drug: Intravenous esketamine using Dixon's up-and-down sequential method — Using Dixon's up-and-down sequential method, esketamine will be titrated intravenously from an initial 0.3 mg∙kg-1 dose with 0.02 mg∙kg-1 adjustments based on intraprocedural responses to pain (Positive: purposeful somatic movement or the complaint of pain; Negative: no movement or no complaint of pain). The titration sequence will continue until six crossover inflection points are observed.
  Other Names: Ultrasound-guided hepatic hilar nerve block (HHNB); Standardized premedication (midazolam 0.03 mg∙kg-1); Local anaesthesia using 10 ml of 1% lidocaine
  Arms: Determine the ED50 and ED95 of esketamine by Dixon's up-and-down method
Drug: Intravenous the dose of esketamine ED95 — The intervention group will be injected with the dose of esketamine ED95.
  Other Names: Ultrasound-guided hepatic hilar nerve block (HHNB); Standardized premedication (midazolam 0.03 mg∙kg-1); Local anaesthesia using 10 ml of 1% lidocaine
  Arms: Evaluate the safety of the dose of esketamine ED95 by the incidence of respiratory depression
Drug: Intravenous fentanyl 1 μg∙kg-1 — The control group will be injected with fentanyl 1 μg∙kg-1.
  Other Names: Ultrasound-guided hepatic hilar nerve block (HHNB); Standardized premedication (midazolam 0.03 mg∙kg-1); Local anaesthesia using 10 ml of 1% lidocaine
  Arms: Evaluate the safety of the dose of esketamine ED95 by the incidence of respiratory depression

SUMMARY:
Effective pain management during percutaneous thermal ablation of liver tumors outside the operating room remains a significant challenge. While hepatic hilar nerve block (HHNB) provides partial analgesia, its incomplete efficacy often requires opioid supplementation, potentially increasing perioperative risks. Esketamine, an N-methyl-D-aspartate receptor antagonist, exhibits unique dual analgesic-sedative properties that may address this therapeutic gap, thus obviating the necessity for opioids. This prospective dose-finding study aimed to establish the median effective dose (ED50) and 95% effective dose (ED95) of esketamine for opioid-free analgesia during ultrasound-guided thermal ablation of liver tumors under HHNB. Afterwards, the investigators will conduct an RCT study to evaluate the safety of the dose of esketamine ED95 through the incidence of respiratory depression.

DETAILED DESCRIPTION:
This research will be divided into two stages.

(i) In Phase one, a prospective dose discovery study using the Dixon sequential method will be conducted, aiming to determine the median effective dose (ED50) and 95% effective dose (ED95) of esketamine during ultrasound-guided thermal ablation of liver tumors under hepatic hilar nerve block (HHNB). Esketamine will be initiated by intravenous drip at 0.3 mg∙kg-1, and then based on the patient's response to pain (positive: body movement or complaint of pain; Negative: No body movement or no reported pain. The dose will be adjusted, with a fluctuation step of 0.02 mg∙kg-1 up and down. All patients will receive a standardized anesthesia regimen, including the administration of midazolam at 0.03 mg∙kg-1 and hepatic portal nerve block (10 ml of 0.5% ropivacaine) under ultrasound guidance. Local anaesthesia will be administered using 10 ml of 1% lidocaine, which will be applied until the liver capsule is reached. The test will continue until six cross-pairings will be obtained. Probabilistic regression analysis will be used to calculate the ED50 and ED95 of esketamine with a 95% confidence interval.

(ii) The investigators will conduct a single-center, randomized, double-blind controlled trial in Phase Two to evaluate the safety of the esketamine ED95 dose under the monitoring anesthesia care program based on the incidence of respiratory depression. The intervention group will be injected with the dose of esketamine ED95; the control group will be first injected with fentanyl at a dose of 1 μg∙kg-1. Both groups of patients will receive the same anesthesia regimen, namely midazolam 0.03 mg∙kg-1, and hepatic portal nerve block (0.5% ropivacaine 10 ml) will be performed under ultrasound guidance. Intravenous injection of 100 mg of flurbiprofen axetil for auxiliary analgesia. Intravenous injection of 4 mg of ondansetron to prevent nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 80 years;
* ASA physical status Ⅰ or Ⅲ;
* Body mass index (BMI) 18 - 28 kg∙m-2;
* Scheduled for elective ultrasound-guided thermal ablation of solitary liver tumors under HHNB.

Exclusion Criteria:

(i) Pharmacological contraindications:

* Known hypersensitivity to study medications (esketamine, midazolam);
* Opioid or benzodiazepine dependence;
* Using analgesics within the last 24 h preoperatively;
* Participation in other investigational drug trials within 90 days. (ii) Clinical comorbidities and surgery history:
* Multifocal hepatic lesions requiring concurrent ablation;
* Patients after liver transplantation;
* Active upper respiratory tract infection within 14 days;
* Severe cardiopulmonary diseases (New York Heart Association [NYHA] class Ⅲ-Ⅳ, FEV1/FVC < 70%);
* Decompensated hepatic insufficiency (Child-Pugh C);
* Uncontrolled hypertension (≥180/110 mmHg), elevated intracranial/intraocular pressure, or hyperthyroidism;
* Major neuropsychiatric disorders (epilepsy, schizophrenia, major depressive disorder, cognitive impairment).

(iii) Procedural Risk Factors:

* Anticipated difficult airway (Mallampati Ⅲ-Ⅳ, thyromental distance < 6 cm) or anatomical airway obstruction;
* Inadequate preoperative fasting (solid intake < 8 hours, clear fluids < 2 hours).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2025-06-29 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
thermal ablation-induced somatic responses to pain | Day 1 (During the surgery at the first stage of the research)
  Positive: Body movement or complaint of pain. Negative: No body movement or no reported pain. This scale will be administered during the surgery at the first stage of the research.
Incidence of respiratory depression | Day 1 (T2-T5 of the second stage of the research)
  By comparing with the control group, evaluate the safety of ED95 of esketamine by the incidence of respiratory depression at T2-T5 of the second stage of the research.
  The primary outcome is the incidence of respiratory depression, which is defined as SpO2 <90% or EtCO2 >55 mmHg.
  T2: 60 seconds after esketamine injection; T3: 5 minutes after HHNB; T4: During thermal ablation of liver tumors; and T5: In the PACU.

SECONDARY OUTCOMES:
HR | Day 1 (T1-T5 of the first and second stages of the research)
  HR: heart rate. T1: Prior to anesthesia (10 minutes after positioning); T2: 60 seconds after esketamine injection; T3: 5 minutes after HHNB; T4: During thermal ablation of liver tumors; and T5: In the PACU.
MAP | Day 1 (T1-T5 of the first and second stages of the research)
  MAP: Mean Arterial Pressure. T1: Prior to anesthesia (10 minutes after positioning); T2: 60 seconds after esketamine injection; T3: 5 minutes after HHNB; T4: During thermal ablation of liver tumors; and T5: In the PACU.
RR | Day 1 (T1-T5 of the first and second stages of the research)
  RR: respiratory rate. T1: Prior to anesthesia (10 minutes after positioning); T2: 60 seconds after esketamine injection; T3: 5 minutes after HHNB; T4: During thermal ablation of liver tumors; and T5: In the PACU.
SPO2 | Day 1 (T1-T5 of the first and second stages of the research)
  SPO2: peripheral oxygen saturation. T1: Prior to anesthesia (10 minutes after positioning); T2: 60 seconds after esketamine injection; T3: 5 minutes after HHNB; T4: During thermal ablation of liver tumors; and T5: In the PACU.
EtCO2 | Day 1 (T2-T5 of the first and second stages of the research)
  EtCO2: End-expiratory carbon dioxide. T2: 60 seconds after esketamine injection; T3: 5 minutes after HHNB; T4: During thermal ablation of liver tumors; and T5: In the PACU.
Adverse events | Day 1 (T2-T8 of the first and second stages of the research)
  Adverse events will encompass a range of systems, including the cardiovascular system (eg. high/low blood pressure and sinus tachycardia/bradycardia), as well as symptoms such as nausea, vomiting, dizziness, and mental symptoms.
  T2: 60 seconds after esketamine injection; T3: 5 minutes after HHNB; T4: During thermal ablation of liver tumors; T5: In the PACU.
  T6 to T8: 2, 6, and 24 hours after the procedure.
NRS | Day 1 (T6-T8 of the first and second stages of the research)
  The Numeric Rating Scale (NRS) will be utilized to assess postoperative pain, with a range of 0 representing no pain and 10 representing severe pain. This scale will be administered at 2, 6, and 24 hours following the procedure.
  T6 to T8: 2, 6, and 24 hours after the procedure.
The need for remedial analgesia | Day 1 (T6-T8 of the first and second stages of the research)
  The consumption of remedial analgesia will be the total consumption of acetaminophen documented at 2, 6, and 24 hours after the procedure.
  T6 to T8: 2, 6, and 24 hours after the procedure.
Success rate of anesthesia | Day 1 (T2-T4 of the second stage of the research)
  Anesthesia success will be defined as inadequate analgesia requiring ≤3 rescue doses of remifentanil within 10 min throughout the procedure. The success rate of anesthesia will be calculated by dividing the number of successful anesthesia cases by the total number of cases.
  T2: 60 seconds after esketamine injection; T3: 5 minutes after HHNB; T4: During thermal ablation of liver tumors
Induction duration | Day 1 of the second stage of the research
  Induction duration is defined as the period from the start of anaesthetic drug injection to the commencement of the surgical procedure at the second stage of the research.
Duration of awakening | Day 1 of the second stage of the research
  Duration of awakening is defined as the period from the conclusion of the surgical procedure to the moment of eye-opening.
Duration of stay in the hospital | Day 1 and Day 2 of the second stage of the research
  Duration of stay in the hospital is measured from the moment the patient enters the operating room until the moment they are discharged.
The satisfaction of the sonographer | Day 1 of the second stage of the research
  The satisfaction score of the sonographer will be collected postoperatively on Day 1, using a scale ranging from 0 to 10, with 0 representing dissatisfaction and 10 representing very satisfied.
The satisfaction of patients | Day 2 of the second stage of the research
  The satisfaction of patients will be collected postoperatively on Day 2, using a scale ranging from 0 to 10, with 0 representing dissatisfaction and 10 representing very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Lijuan Yan, Principal Investigator — Department of Anesthesiology, The First Affiliated Hospital of Xiamen University
Locations (1):
- Department of Anesthesiology, The First Affiliated Hospital of Xiamen University, 55 Zhenhai Road, Xiamen, China, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No